CLINICAL TRIAL: NCT07378085
Title: The Impact of Virtual Reality Games on Upper Extremity Function, Activity, and Participation in Hemiplegic Patients: A Randomized Controlled Trial
Brief Title: Virtual Reality-Based Upper Limb Rehabilitation in Hemiplegia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Principal Investigator, Pinar Dogan, Medical doctor, Gaziosmanpasa Research and Education Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 07
Record Dates: First submitted 2025-12-10; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-12

CONDITIONS: Upper Extremity Hemiplegia; Stroke; Virtual Reality Based Therapy
Keywords: stroke rehabilitation; virtual reality; upper extremity; motor skills; leap motion
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: The study is a single-blind, prospective, randomized controlled, single-center study. Patients were randomly assigned to the experimental group (EG) or the control group (CG). A box containing 40 opaque, sealed envelopes was prepared: 20 labeled "CG" and 20 "EG". Occupational therapists asked participants to draw one envelope. If they withdrew from the study, the envelope corresponding to their group was returned. The study continued until all 40 envelopes had been drawn and complete data were collected.
Who Masked: Outcomes Assessor
Masking Description: The study was conducted in a single-blind manner, only the evaluator did not know which patient was in the experimental group and which patient was in the control group. Due to the nature of the treatment, the patients and the occupational therapist performing the game were not blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): The control group received conventional rehabilitation for 1 hour every day, 5 days a week for 4 weeks.
  Interventions: Other: conventional rehabilitation
- experimental group (Active Comparator): In addition to conventional rehabilitation, participants in the experimental group received Leap Motion-based virtual reality therapy 5 days per week for 4 weeks. For this purpose, the Leap Motion device, leased from Becure GmbH (GOSB Teknopark Hightech Building, Gebze, Kocaeli, Turkey), was used to deliver a computer-based HandROM program designed to improve upper extremity functions. Each session consisted of 4 games, played for 10 minutes each, resulting in a total of 40 minutes of additional upper extremity exercise per day. Four therapeutic games used in intervention are as follows: Leap Maze, Leap Ball , Pong and CatchAPet. During the games, patients performed forearm pronation-supination, wrist flexion-extension, and finger flexion-extension movements.
  Interventions: Other: conventional rehabilitation; Device: leap motion based virtual reality rehabilitation

INTERVENTIONS:
Other: conventional rehabilitation — Conventional rehabilitation consisted of joint range of motion exercises, stretching, strengthening, balance and postural control training, transfer training, gait training, stair climbing exercises, and neurophysiological exercise techniques, all performed under the supervision of a physiotherapist.
Device: leap motion based virtual reality rehabilitation — The VR system was implemented using the Leap Motion device, which incorporates an infrared depth sensor capable of detecting limb movements in three-dimensional space. This technology enables users to interact with the virtual environment without the need for a handheld controller; instead, the user's upper extremities function directly as the interface. During the intervention, patients participated in computer-based rehabilitation while seated, with the motion sensor positioned to accurately capture hand and wrist movements.
  Arms: experimental group

SUMMARY:
This study aims to evaluate the effectiveness of Leap Motion-supported virtual reality therapy, applied in addition to traditional rehabilitation programs, in individuals who develop hemiplegia after a cerebrovascular accident. The study will examine the effects of this additional therapy on upper extremity functions, activities of daily living, and participation levels.

DETAILED DESCRIPTION:
Hemiplegic patients experience significant limitations in their activities of daily living (ADL) and participation levels due to marked losses in upper extremity function following stroke. Approximately 80% of individuals who have had a stroke experience impairment in upper extremity function, and because the upper extremity plays a critical role in many motor functions, these impairments significantly affect independence. Therefore, initiating upper extremity rehabilitation early and tailoring it to the individual's needs is of great importance for functional improvement. Various treatment methods are used in stroke rehabilitation to support physical, functional, and psychological recovery.

In recent years, virtual reality-based technologies have been increasingly used in rehabilitation processes due to their ability to increase motivation, enable intensive and repetitive motor training, and provide environmental feedback. Leap Motion-based virtual reality applications enable patients to participate in therapy through safe, interactive, and task-oriented activities by allowing three-dimensional perception of upper extremity movements.

The aim of this study is to compare the effects of Leap Motion-based virtual reality rehabilitation, applied in addition to conventional treatment, on the functional development of the plegic upper extremity, activities of daily living, and participation levels compared to the group receiving conventional treatment alone.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be above eighteen years of age
* Have had a first-time stroke
* Be within twelve months of stroke
* Have a Brunnstrom score of four or more for the upper extremity
* Be cognitively adequate (scoring ≥23 on the mini-mental test scale)

Exclusion Criteria:

* Being in the unstable phase of the disease
* Visual and/or auditory impairments
* Unilateral spatial neglect (hemineglect)
* Modified Ashworth Scale score of ≥3 in the affected upper limb
* Had a history of botulinum toxin A (Botox) injection in the affected upper limb within the previous six months
* Other systemic neuromuscular disorders (exc; Alzheimer Disease, Parkinson Disease, Multipl Sclerosis...)
* Have cerebellar involvement characterised by dysmetria, dysdiadochokinesia or ataxia
* Have a prior orthopaedic or neuromuscular injuries affecting both upper limbs
* Have impaired static sitting balance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-01-23 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer assessment for upper extremity | baseline (T0), at the end of treatment (T1), one month after treatment completion (T2), and three months after treatment completion (T3)
  In our study, we used the upper extremity motor evaluation part of the Fugl-Meyer scale. This scale is valid and reliable in evaluating motor recovery after stroke. This scale has 4 subheadings: arm evaluation (maximum 36 points), wrist evaluation (10 points), hand evaluation (maximum 14 points), coordination and speed (maximum 6 points). It consists of 33 items scored from 0 to 2. '0: Cannot realize, 1: Partially realizes, 2: Completely realizes'. A maximum of 66 points can be obtained in the upper extremity scoring. Higher scores indicate better motor recovery.

SECONDARY OUTCOMES:
Selective Control of the Upper Extremity Scale | baseline (T0), at the end of treatment (T1), one month after treatment completion (T2), and three months after treatment completion (T3)
  It evaluates selective movements in the shoulder, elbow, forearm, wrist and fingers. The person to be evaluated is seated at a table wearing appropriate clothing so that his or her extremities can be clearly seen. The assessor himself shows how to perform the movements. Then the participant actively performs the movement. While the participant is performing the movements, the movements of the head, trunk and both extremities are recorded on a video camera so that they are fully visible. Scoring for each joint is "Normal Selective Motor Control" (3 points), "Mildly Decreased Selective Motor Control" (2 points), "Moderately Decreased Selective Motor Control" (1 point), and "No Selective Motor Control" (0 points). score). A maximum of 15 points can be obtained for the extremity evaluated. A higher score indicates better selective motor control in that limb.
Stroke Specific Quality of Life Scale | baseline (T0), at the end of treatment (T1), one month after treatment completion (T2), and three months after treatment completion (T3)
  It is used to evaluate quality of life after stroke. SS-QOL consists of 12 subsections (mobility (6 items), energy (3 items), upper extremity function (5 items), work/production (3 items), temperament (5 items), self-care (5 items), social role (5 items). item), family role (3 items), vision (3 items), language (5 items), thinking (3 items) and personality traits (3 items) and a total of 49 questions. Each question was rated with a Likert-type score ranging from 1 to 5. Rating "1. "I couldn't do it at all, 2. I found it very difficult, 3. I found it a little difficult, 4. I found it very little difficult, 5. I did not find it difficult at all." A maximum of 245 points can be obtained. A high scale score indicates a high quality of life, and a low scale score indicates a low quality of life.
Turkish Version of Disabilities of The Arm, Shoulder and Hand | baseline (T0), at the end of treatment (T1), one month after treatment completion (T2), and three months after treatment completion (T3)
  This questionnaire was developed to evaluate the functional status and ability to perform activities of daily living in patients with upper extremity injuries. In our study, the first part of the DASH-T survey, consisting of 30 questions, was applied. Of these 30 questions, 21 evaluate the person's difficulties during daily living activities, 5 evaluate the symptoms (pain, stiffness, tingling, weakness), and 4 evaluate work, sleep, social function and self-confidence. The person answers all questions according to a 5-point Likert system (1: no difficulty, 2: mild difficulty, 3: moderate difficulty, 4: extreme difficulty, 5: not able to do it at all). When calculating the total score, the total score of the marked items is divided by the number of marked items and subtracted by 1. The result is then multiplied by 25. A score between 0-100 is obtained. As the score increases, the disability also increases.
nine hole peg test | baseline (T0), at the end of treatment (T1), one month after treatment completion (T2), and three months after treatment completion (T3)
  The Nine-Hole Peg Test (NHPT) is a simple test of manual dexterity. It assesses fine motor coordination and finger-hand speed. Participants pick up nine pegs from a container, one by one, and insert them into the holes on a pegboard as quickly as possible. Participants must remove pegs one by one and return them to the container after inserting them. The stopwatch records the time taken. Longer times indicate poorer manual dexterity

CONTACTS AND LOCATIONS:
Overall Officials: Pinar Dogan, MD, Principal Investigator — Gaziosmanpasa Research and Education Hospital
Locations (1):
- Gaziosmanpasa Research and Education Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The data obtained from patients participating in the statistical analysis will be shared without disclosing patient identities.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After the study results are published, these data will be made available for use. Study data can be shared for one year
Access Criteria: Upon request, and subject to ethical approval or data usage agreements, the data will be shared with qualified researchers affiliated with academic or medical institutions. Data can be obtained by Principal Investigator Email Address: pinar.karagoz94@gmail.com

REFERENCES:
- [Background] Ogun MN, Kurul R, Yasar MF, Turkoglu SA, Avci S, Yildiz N. Effect of Leap Motion-based 3D Immersive Virtual Reality Usage on Upper Extremity Function in Ischemic Stroke Patients. Arq Neuropsiquiatr. 2019 Oct 24;77(10):681-688. doi: 10.1590/0004-282X20190129. eCollection 2019. PMID 31664343
- [Background] Wang ZR, Wang P, Xing L, Mei LP, Zhao J, Zhang T. Leap Motion-based virtual reality training for improving motor functional recovery of upper limbs and neural reorganization in subacute stroke patients. Neural Regen Res. 2017 Nov;12(11):1823-1831. doi: 10.4103/1673-5374.219043. PMID 29239328
- [Background] Shin JH, Kim MY, Lee JY, Jeon YJ, Kim S, Lee S, Seo B, Choi Y. Effects of virtual reality-based rehabilitation on distal upper extremity function and health-related quality of life: a single-blinded, randomized controlled trial. J Neuroeng Rehabil. 2016 Feb 24;13:17. doi: 10.1186/s12984-016-0125-x. PMID 26911438